CLINICAL TRIAL: NCT06698796
Title: A PHASE 3, MULTI-CENTER, OPEN-LABEL EXTENSION STUDY TO INVESTIGATE THE LONG-TERM SAFETY, TOLERABILITY, AND EFFICACY OF DAZUKIBART IN PARTICIPANTS WITH IDIOPATHIC INFLAMMATORY MYOPATHIES (INCLUDING PARTICIPANTS WITH DERMATOMYOSITIS OR POLYMYOSITIS)
Brief Title: A Study to Understand How the Study Medicine Dazukibart Works in People With Idiopathic Inflammatory Myopathies
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C0251010; 2024-514648-10-00 (Registry Identifier: CTIS (EU))
Expanded Access: Available
Record Dates: First submitted 2024-10-24; First posted 2024-11-21 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Dermatomyositis; Polymyositis
MeSH Terms: conditions — Dermatomyositis; Polymyositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dazukibart (Experimental): Participants will receive dazukibart via intravenous infusion every 4 weeks.
  Interventions: Drug: Dazukibart

INTERVENTIONS:
Drug: Dazukibart — anti-interferon beta therapy

SUMMARY:
The purpose of this study is to understand how the study medicine, dazukibart, works in people with active idiopathic inflammatory myopathies (dermatomyositis [DM] or polymyositis [PM]).

Idiopathic inflammatory myopathies are a group of disorders that show inflammation of the muscles used for movement. There are several types of idiopathic inflammatory myopathies, including DM and PM.

DM and PM involve weakness of the muscles closest to the center of the body, such as the muscles of the hips, thighs, upper arms, and neck. People with these forms of idiopathic inflammatory myopathies may find it difficult to climb stairs, get up from a seated position, or lift items above their head. People with DM can also have a skin rash.

These disorders negatively impact the quality of life and functioning of patients. In addition to the above, these disorders can affect how the lungs and heart work.

This study is seeking participants who took part in a DM and PM study with dazukibart before. Some participants will receive study medicine, and some participants will not receive study medicine and only complete safety follow-up.

The study medicine will be given as an intravenous (IV) infusion (directly into the veins). This takes about 1 hour, every 4 weeks, from Day 1 to Week 48 (about 12 months) of the study. This will be followed by a safety follow-up period that lasts about 4 months after the last infusion. Participants who receive study medicine will have about 18 study visits at the site over about 16 months.

There will also be participants enrolled in this study who will not receive study medicine. Such participants will only take part in safety follow-up visits as they do not want to or are not eligible to receive dazukibart. These participants will not receive study medicine and will have up to 4 study visits at the site every 4 weeks to complete safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants that completed a qualifying study through Week 52.

Exclusion Criteria:

* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation.
* Previous administration with an investigational product (drug or vaccine) other than dazukibart in a qualifying study within 30 days (or as determined by the local requirement) or 5 half-lives preceding baseline in this study (whichever is longer).
* Current use of any prohibited concomitant medication(s).
* Active bacterial, viral, fungal, mycobacterial or other infections.
* Ongoing adverse event in a qualifying study or the participant has met safety monitoring criteria in a qualifying study that have not resolved.
* Investigator site staff or sponsor employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2027-11-25 (Estimated); Study Completion 2027-11-25 (Estimated)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events (AEs), Serious AEs, AEs of Special Interest, and AEs leading to treatment discontinuation | 52 weeks
  An AE is any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. Treatment-emergent are AEs that are absent before treatment or that worsened relative to pretreatment state. Pre-defined AESI for this study are outlined in study protocol.
Number of participants with clinically significant laboratory abnormalities | 52 weeks
  Clinically significant laboratory abnormalities are those that meet the Common Terminology Criteria for Adverse Events (CTCAE) definition.
Number of participants with clinically significant abnormalities in vital signs | 52 weeks
  Clinically significant vital sign abnormalities include pulse rate <40, >100 or >120 bpm; systolic blood pressure increase from baseline ≥30 or decrease ≤30 mmHg; diastolic blood pressure increase from baseline ≥20 or decrease ≤20 mmHg.
Number of participants with clinically significant electrocardiogram (ECG) abnormalities | 52 weeks
  Clinically significant ECG abnormalities include mild (>450-480 millisecond [msec]), moderate (>480-500 msec or 30-60 msec increase from baseline), and severe (>500 msec or >60 msec increase from baseline) QTc prolongation.
Change from baseline in Forced Vital Capacity (FVC)/Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) | 52 weeks
  FVC is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. DLCO is a measure of gas exchange diffusion capacity.
Absolute values and change from baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) | 52 weeks
  C-SSRS assesses whether participant experienced following: completed suicide (1), suicide attempt (2) (response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3)("Yes" on "preparatory acts or behavior"), suicidal ideation (4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior (7)("Yes" on "Has subject engaged in non-suicidal self-injurious behavior").

SECONDARY OUTCOMES:
Change from baseline in Manual Muscle Testing - 8 designated muscles (MMT-8) | 52 weeks
  Manual Muscle Testing (8 designated muscles) 0 to 150 with higher scores indicating a better outcome
Change from baseline in Physician Global Activity (PhGA) | 52 weeks
  Physician Global Activity 0 to 10 scale with higher scores indicating a worse outcome
Change from baseline in extramuscular activity or disease activity score and muscle enzyme results | 52 weeks
  Results come from Total Improvement Score 0 to 100 with higher scores indicating a better outcome and laboratory values
Minimal, Moderate, and Major improvement in Total Improvement Score (TIS) and TIS (continuous) score | 52 weeks
  Total Improvement Score 0 to 100 with higher scores indicating a better outcome.
Percent change from baseline and change from baseline in Cutaneous Dermatomyositis Disease Area and Severity Index Activity Score (CDASI-A) in DM participants | 52 weeks
  Cutaneous Dermatomyositis Disease Area and Severity Index Activity Score 0 to 100 with higher scores indicating a worse outcome
Change from baseline in Cutaneous Dermatomyositis Disease Area and Severity Index Damage Score (CDASI-D) in DM participants | 52 weeks
  Cutaneous Dermatomyositis Disease Area and Severity Index Damage Score 0 to 32 with higher scores indicating a worse outcome
Change from baseline in Patient-Reported Outcomes Measurement Information System - Physical Function (PROMIS-PF) | 52 weeks
  Patient-Reported Outcomes Measurement Information System - Physical Function 0 to 100 with higher scores indicating a better outcome
Change from baseline in Patient Global Activity (PtGA) | 52 weeks
  Patient Global Activity 10-point numeric rating scale with higher scores indicating worse outcome
Change from baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) | 52 weeks
  Health Assessment Questionnaire-Disability Index 20 questions with 0 to 3 scale where higher scores indicate a worse outcome
Change from baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | 52 weeks
  Functional Assessment of Chronic Illness Therapy - Fatigue 0 to 52 with higher scores indicating a better outcome
Change from baseline in EuroQoL 5 Dimensions (EQ-5D-5L) and EuroQoL Visual Analog Scale (EQ-VAS) | 52 Weeks
  EuroQoL 5 Dimensions and EuroQoL Visual Analog Scale with higher scores indicating a worse outcome
Change from baseline in Healthcare Resource Utilization Questionnaire (HRU) | 52 weeks
  Healthcare Resource Utilization Questionnaire measures the healthcare utilization burden while on treatment
Change from baseline in 5-D Itch Scale Score in DM participants | 52 weeks
  5-D Pruritis Scale 5 to 25 with higher scores indicating a worse outcome
Change from baseline in corticosteroid (CS) and non-steroid immunosuppressant/immunomodulator and antimalarial dose | 52 weeks
  CS and non-steroid immunosuppressant/immunomodulator and antimalarial dose
Response in CS and non-steroid immunosuppressant/immunomodulator and antimalarial tapering | 52 weeks
  CS dose ≤5 mg/day or CS and non-steroid immunosuppressant/immunomodulator and antimalarial free
Rescue therapy use assessment | 52 weeks
  Rescue therapy received during the study and number of cycles
Auto antibodies and immunogenicity presence | 52 weeks
  Auto antibody lab assessment (eg. TIF1-γ/P155, NXP2/P140, SAE, JO-1 and MDA-5) and ADAs/Nabs

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (2):
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Glendale, Glendale, Arizona
  - Rheumatology & Pulmonary Clinic, Beckley, West Virginia
- Medical Center Artmed, Plovdiv, Bulgaria
- China (3):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Renji Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
- CHARM HEALTHCARE PRIVATE LIMITED (Previously Dr Shenoy's Care Private Limited), Ernākulam, Kerala, India
- Japan (2):
  - Institute of Science Tokyo Hospital, Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0251010